CLINICAL TRIAL: NCT06661447
Title: Comparison of Bone Augmentation Techniques in the Mandible Posterior Region: a Randomized Split-mouth Trial
Brief Title: Bone Augmentation Techniques in the Mandible Posterior Region
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Especialidades Espiritu Santo (Other)
Responsible Party: Principal Investigator, Antonio Lanata Flores, Assistant Professor, Universidad de Especialidades Espiritu Santo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-ODONT-002
Record Dates: First submitted 2024-09-02; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Bone Substitutes; Alveolar Bone Grafting
Keywords: Alveolar Bone Atrophy; Bone Substitutes; Bone Resorption
MeSH Terms: conditions — Alveolar Bone Loss; Bone Resorption

STUDY DESIGN:
Intervention Model Description: Split mouth randomized clinical trial will performed in 40 patient with bilateral edentulous atrophic posterior region.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants will not know which technique is being used in their edentulous area.
  The investigator will not be informed which grafting technique was performed in the edentulous areas.
  The outcomes assessor will not be informed of which procedures were performed on the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Autogenous Onlay bone graft (Active Comparator): All patients will be submitted under a Onlay bone graft Technique with autogenous block bones is perform in one of the two Bilateral Mandibular Posterior Edentulous areas. The inner space is filled with a mixture of autogenous and xenogeneic particulated bone
  Interventions: Procedure: Tridimensional Onlay autologous bone graft
- Xenogeneic Onlay bone graft (Experimental): In 20 patients, A xenogeneic onlay bone graft is positioned in the remaining mandibular posterior edentulous area. The inner space is filled with a mixture of autogenous and xenogeneic particulated bone
  Interventions: Procedure: Tridimensional Onlay xenogeneic bone graft
- Allogenic Onlay bone graft (Experimental): In 20 patients, A allogenic onlay bone graft is positioned in the remaining mandibular posterior edentulous area. The inner space is filled with a mixture of autogenous and xenogeneic particulated bone
  Interventions: Procedure: Tridimensional Onlay allogenic bone graft

INTERVENTIONS:
Procedure: Tridimensional Onlay autologous bone graft — A thick block from the ramus area of the mandible are cut longitudinally with a microsaw into two thin pieces with the same surface area. The two thin block are used to rebuild the two wall of the future alveolar crest and stabilized with osteosynthesis screw of the edentulous area. The remaining space is filled with a mixture of autogenic and xenogeneic particulate bone.
  Other Names: Shell technique; 3D Onlay bone graft; Khoury´s bone graft technique
  Arms: Autogenous Onlay bone graft
Procedure: Tridimensional Onlay xenogeneic bone graft — A tridimensional Onlay xenogeneic bone graft is positioned and stabilized with osteosynthesis screw of the edentulous area. The remaining space is filled with a mixture of autogenic and xenogeneic particulate bone.
  Arms: Xenogeneic Onlay bone graft
Procedure: Tridimensional Onlay allogenic bone graft — A tridimensional Onlay allogenic bone graft is positioned and stabilized with osteosynthesis screw of the edentulous area. The remaining space is filled with a mixture of autogenic and xenogeneic particulate bone.
  Arms: Allogenic Onlay bone graft

SUMMARY:
This study aims to compare the efficacy of two bone augmentation techniques in the posterior mandible. Twenty participants will undergo 40 surgical procedures at Espíritu Santo University (UEES) in Samborondon, Ecuador. Each patient will receive two types of bone grafts: one side will use autogenous cortical bone plates with a 50/50 mixture of autogenous bone and biomaterial (as described by Dr. Fouad Khoury), while the other side will use xenogenous cortical bone plates with the same mixture.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Bilateral Mandibular Posterior Edentulous with atrophy in 4, 5 or 6 Cawood and Howell stages.
* Patients who have good plaque control of less than 20%
* Patients between 18-64 years old

Exclusion Criteria:

* Systemically compromised patients
* Smoker patients
* Pregnant women, breastfeeding or use of oral contraceptives
* Patients who are taking medication that may affect healing and coagulation
* Patients with periodontal disease
* Patients who have undergone chemotherapy and radiotherapy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2029-12-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate bone formation Across Different Graft Techniques | The evaluation will occur from enrollment through the end of treatment at 12 months. Assessments will be conducted preoperatively, 7 days post-surgery, as well as at 3, 6, and 12 months following the surgery.
  This study aims to evaluate bone formation resulting from various bone grafting techniques, with a focus on quantifying the amount of newly formed bone.

SECONDARY OUTCOMES:
To evaluate the surgery duration of across different bone grafting techniques. | To record the duration of surgery for both techniques, from the administration of anesthesia to the final suture
  This study aims to evaluate the surgery duration.
To evaluate bone quality across different bone grafting techniques. | From enrollment, to the end of treatment at 12 months; evaluating at 3 days, 30 days, 3 months, 6 months and 12 months
  This will involve analyzing the bone density through radiographic imaging.
To evaluate postoperative inflammation across different bone grafting techniques. | The evaluation will occur prior to surgery, immediately postoperatively, on the 3rd day, 7th day, and at 14 days
  This study aims to evaluate postoperative inflammation following surgery. A measurement will be taken from the corner of the lip to the ear lobe using a flexible measuring tape in order to monitor the swelling. The data will be recorded in millimeters.

REFERENCES:
- [Background] Khoury F, Hanser T. Three-Dimensional Vertical Alveolar Ridge Augmentation in the Posterior Maxilla: A 10-year Clinical Study. Int J Oral Maxillofac Implants. 2019 Mar/Apr;34(2):471-480. doi: 10.11607/jomi.6869. PMID 30883623